CLINICAL TRIAL: NCT06766357
Title: A Phase 3, Multicenter, Randomized, Double-blind, Vehicle-controlled Efficacy and Safety Study of Cyclosporin Ophthalmic Gel in Subjects With Moderate to Severe Dry Eye Disease
Brief Title: A Study of the Efficacy and Safety of Cyclosporin Ophthalmic Gel in Subjects With Moderate to Severe Dry Eye Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKO-CSP-CSA-302
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-01

CONDITIONS: Moderate to Severe Dry Eye
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): 1 drop each time, once every night at bedtime
  Interventions: Drug: Cyclosporine ophthalmic gel
- Control group (Placebo Comparator): 1 drop each time, once every night at bedtime
  Interventions: Drug: Cyclosporine ophthalmic gel vehicle

INTERVENTIONS:
Drug: Cyclosporine ophthalmic gel — Administer to eyes
  Other Names: Cyclosporine
  Arms: Experimental group
Drug: Cyclosporine ophthalmic gel vehicle — Administer to eyes
  Other Names: Vehicle
  Arms: Control group

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled, superiority design Phase III clinical trial. The primary objective is to evaluate the efficacy and safety of cyclosporine ophthalmic gel versus placebo in the treatment of moderate to severe dry eye for 84 days.

DETAILED DESCRIPTION:
A total of 360 subjects are planned to be enrolled in this study. This study is divided into two stages. The first stage (double-blind treatment period) is the main efficacy and safety evaluation stage, which lasts for 84 days. During this period, subjects are randomly assigned to receive the experimental drug or control drug in a 1:1 ratio, with the analysis of the first stage as the main analysis. After completing the 84th day visit, the subjects will enter the second stage (open treatment period). The second stage is a safety observation period of 84 days, during which all subjects use the experimental drug.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 18 years old, males or females.
2. Subjects complained of ocular dryness in both eyes for at least 6 months at Visit 1.
3. Eye dryness score(EDS)(evaluated on a 0-100 VAS score) ≥40 at Visit 1 and Visit 2.
4. Ocular Surface Disease Index (OSDI) score ≥13 at Visit 1 and Visit 2.
5. Total corneal fluorescein staining score (tCFS) ≥2 in either eye and ≥1 in at least one region at Visit 1 and Visit 2.
6. Schirmer I test (without anesthesia) ≤ 5 mm/5 min in either eye at Visit 1 and Visit 2.
7. Subjects with moderate and severe dry eye in both eyes at Visit 1 and Visit 2:

   1. Moderate: ≥1 quadrant and no more than 2 quadrants of corneal damage and/or ≥5 and <30 corneal fluorescein staining spots on slit lamp microscopy;
   2. Severe: ≥2 quadrants of corneal damage and/or ≥30 corneal fluorescence staining spots on slit lamp microscopy.

Exclusion Criteria:

1. Subjects with severe dry eye requiring surgical treatment.
2. Systemic use of retinoids within the 12 months prior to Visit 1.
3. Subjects who have had intraocular surgery within 12 months prior to Visit 1 or who require intraocular surgery during the study; or subjects who have had eyelid surgery within 6 months prior to Visit 1.
4. Subjects treated with permanent lacrimal duct embolization; or subjects treated with temporary lacrimal duct embolization within 6 months prior to Visit 1.
5. Subjects with dry eye correlated with operation；
6. Subjects who had worn corneal contact lens within 3 months prior to Visit 1.
7. Those who have used cyclosporine preparations ocularly or systemically within 1 month prior to visit 1.
8. Those who have used lifitegrast eye drops or tacrolimus eye drops ocularly within 1 month prior to visit 1.
9. Subjects with dry eye secondary to scarring (e.g., radiation exposure, ocular chemical burns, Stevens-Johnson syndrome, keloid pemphigoid, conjunctival scarring) or severe conjunctival cup cells destruction (e.g., vitamin A deficiency).
10. Those with significant eyelid margin inflammation or meibomian gland dysfunction that, in the opinion of the investigator, may affect the outcome of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Eye Dryness Score(EDS) | 84 days
  Mean change from baseline in EDS scores (evaluated on a 0-100 VAS score) on Day 84 (binocular)

SECONDARY OUTCOMES:
Eye Dryness Score(EDS) | 14 days and 42 days
  Mean change from baseline in EDS scores (evaluated on a 0-100 VAS score) on Day 14 and Day 42 (binocular)
Total VAS score for dry eye symptoms | 14 days, 42 days and 84 days
  Mean change from baseline in total VAS score of dry eye symptoms (evaluated on a 0-100 VAS score) on Day 14, Day 42 and Day 84 (binocular)
Total corneal fluorescein staining score(tCFS) | 14 days, 42 days and 84 days
  The proportion of subjects with a total corneal fluorescein staining score (tCFS, modified NEI scale) of 0 on Day 14, Day 42, and Day 84 (study eye)
Schirmer test | 14 days, 42 days and 84 days
  The proportion of subjects with a change of ≥ 10mm from baseline in the Schirmer test (tear secretion test) on Day 14, Day 42, and Day 84 (study eye)
tear film break-up time(BUT) | 14 days, 42 days and 84 days
  Mean change from baseline in tear film break-up time (BUT) measurements on Day 14, Day 42, and Day 84 (study eye)

CONTACTS AND LOCATIONS:
Overall Officials: Zuguo Liu, Principal Investigator — Xiamen Eye Center of Xiamen University
Locations (1):
- Xiamen Eye Center of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No